CLINICAL TRIAL: NCT02582008
Title: Smoking Cessation in Patients With Squamous Cell Cancer of the Head and Neck Undergoing Radiation Therapy With or Without Chemotherapy
Brief Title: Bupropion Hydrochloride or Patient's Choice for Smoking Cessation in Patients With Squamous Cell Head and Neck Cancer Undergoing Radiation Therapy With or Without Chemotherapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00035113; NCI-2015-01714 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU # 98415; CCCWFU 98415 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2021-06

CONDITIONS: Current Smoker; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Nasopharyngeal Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma | interventions — Bupropion; Nicotine Replacement Therapy; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (bupropion hydrochloride) (Experimental): Patients receive bupropion hydrochloride PO for 3 days and then BID for up to 1 year post RT/CRT.
  Interventions: Drug: Bupropion Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (varenicline, NRT) (Active Comparator): Patients receive smoking cessation treatment tailored to individual smokers based on preference, smoking history and contra-indications. Patients are given the choice of one of the NCCN-recommended first-line pharmacotherapy options for smoking cessation comprised of varenicline PO daily for 1 week and then BID for 12 weeks or combination of nicotine patch and acute NRT for 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Treatment with varenicline or NRT can be extended up to 6 months to 1 year as needed.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nicotine Replacement; Other: Questionnaire Administration; Drug: Varenicline

INTERVENTIONS:
Drug: Bupropion Hydrochloride — Given PO
  Other Names: Amfebutamone; BW 323U66; Forfivo XL; Wellbutrin; Zyban
  Arms: Arm A (bupropion hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nicotine Replacement — Given NRT
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm B (varenicline, NRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm A (bupropion hydrochloride)
Other: Questionnaire Administration — Ancillary studies
Drug: Varenicline — Given PO
  Other Names: Champix; Chantix; CP-526555
  Arms: Arm B (varenicline, NRT)

SUMMARY:
This pilot randomized clinical trial studies how well bupropion hydrochloride works compared with patient's choice for quitting smoking in patients with squamous cell head and neck cancer undergoing radiation therapy with or without chemotherapy. Bupropion hydrochloride may help patients quit smoking by enhancing central nervous system neurotransmitters noradrenergic and dopaminergic release. It is not yet known whether bupropion hydrochloride is more effective than patient's choice in helping quit smoking in patients with squamous cell head and neck cancer undergoing radiation therapy with or without chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who are not smoking (successful quitters) at 12 months post-radiation therapy (RT)/chemotherapy and radiation therapy (CRT) and compare proportions between the two study arms.

SECONDARY OBJECTIVES:

I. To compare the proportion of patients who are not smoking at 6 months post-RT/CRT between the two study arms.

II. Among patients who quit smoking, determine the proportion of patients who experience smoking relapse at 12 months post-RT/CRT and compare between the two study arms.

III. To compare the maximum degree of mucositis and mucositis-related pain during radiation treatment and the following week post-treatment between the two study arms.

IV. Determine the impact of study treatment on anxiety, depression and quality of life (QOL) and compare between two study arms.

V. Collect descriptive data assessing smoking status among caregivers and corresponding data concerning whether smoking relapse occurs in our patient population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive bupropion hydrochloride orally (PO) for 3 days and then twice daily (BID) for up to 1 year post RT/CRT.

ARM B: Patients receive smoking cessation treatment tailored to individual smokers based on preference, smoking history and contra-indications. Patients are given the choice of one of the National Comprehensive Cancer Network (NCCN)-recommended first-line pharmacotherapy options for smoking cessation comprised of varenicline PO daily for 1 week and then BID for 12 weeks or combination of nicotine patch and acute nicotine replacement therapy (NRT) for 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Treatment with varenicline or NRT can be extended up to 6 months to 1 year as needed.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell carcinoma of the nasopharynx, oropharynx, larynx, hypopharynx, oral cavity
* Patients must be scheduled to receive RT or CRT as definitive treatment or surgery with planned adjuvant RT or CRT treatment post-surgery per surgeon or Head and Neck Cancer (HNC) Tumor Board decision
* Patients should receive their definitive treatment at Wake Forest University (WFU) Cancer Center or at Medical University of South Carolina (MUSC) Cancer Center
* Patients must be active smokers (defined as smoking any cigarette, cigar or pipe in the last 30 days)
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients who receive RT or CRT with palliative intent and have a prognosis of less than one year survival
* Patients who chew tobacco and patients who are not smoking but are exposed to second hand smoking are excluded from this study
* Patients currently using a smoking cessation treatment
* Other known drug use/abuse
* Patients with documented contraindications for bupropion (bupropion hydrochloride), including: bulimia nervosa, anorexia nervosa; use of monoamine oxidase inhibitors in the past two weeks; documented seizure disorders or predisposition to seizure (ie stroke, brain metastases); abrupt withdrawal from alcohol, benzodiazepines, or other sedatives; closed-angle glaucoma
* Patients with diagnosis of major depression or any other psychiatric disorders
* Documented history of allergic reactions attributed to compounds of similar chemical or biologic composition to buproprion
* Any other significant acute or chronic diseases that in the investigator's opinion would exclude the subject from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are not smoking | At 12 months post RT or CRT
  Observed rates of patients who are not smoking at 12 months and corresponding 95% exact Clopper-Pearson confidence intervals will be estimated. Next, will perform a Fisher's exact test to determine whether the proportion of patients who are not smoking at 12 months post-RT/CRT in the bupropion hydrochloride group and the patient's choice group are different.

SECONDARY OUTCOMES:
Levels of depression and anxiety as measured by Hamilton Rating Scale-Depression questionnaire | Up to 12 months
  Compared using two sample t-tests.
Proportion of patients who are not smoking at 6 months post RT or CRT | At 6 months
  Study arms will be compared using Fisher's exact tests. Proportions and 95% exact Clopper Pearson confidence intervals will be estimated for each group as well.
Proportion of patients who develop mucositis and mucositis-related pain evaluated by Common Terminology Criteria for Adverse Events | Up to 2 weeks post RT or CRT
  This will be examined by treatment group. Within each group will examine the proportion, confidence interval and also the distribution of grade for these measures.
Proportion of patients who experience smoking relapse among patients who quit smoking | At 12 months post RT or CRT
  This proportion will be calculated for each group and 95% exact Clopper-Pearson confidence intervals will be estimated. The groups will then be compared using a Fisher's exact test.
QOL as measured by MD Anderson Inventory | Up to 12 months
  Compared using two sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440

DOCUMENTS (1):
  • Informed Consent Form (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT02582008/ICF_000.pdf